CLINICAL TRIAL: NCT01790776
Title: Diagnosis of Urethral Stricture With Sono-urethrography vs Conventional Urethrography: Evaluation of the Diagnostic Value and Evaluation of the Reduction of the Radiation Dose With Sono-urethrography (SONO-URETHRA)
Brief Title: Diagnosis of Urethral Stricture With Sono-urethrography vs Conventional Urethrography (SONO-URETHRA)
Acronym: SONO-URETHRA
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2012/902
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Urethral Stricture Disease
Keywords: urethrography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional urethrography (Active Comparator): Current golden standard.
  Interventions: Radiation: Urografin 30%
- Sono-urethrography (Experimental): Experimental urethrography, which could be followed by conventional urethrography if the results are inconclusive.
  Interventions: Radiation: NaCl 0,9 % in aqua

INTERVENTIONS:
Radiation: Urografin 30% — Urografin 30% (Natrium amidotrizoas 10G, Megalumin, Amidotrizoas 65G, Natrii calcii edetas, water for injection 250 ml, with 146 mg iodium/ml).
  The tip of a bladder catheter is placed at the external urethral meatus and fixed at this location. The solution (urografin 30 %) is instilled.
  Arms: Conventional urethrography
Radiation: NaCl 0,9 % in aqua — The tip of a bladder catheter is placed at the external urethral meatus and fixed at this location. The solution (NaCl 0,9 % in aqua) is instilled. If the result is inconclusive, urografin 30 % will be instilled.
  Arms: Sono-urethrography

SUMMARY:
Conventional urethrography is the standard diagnostic evaluation for patients with a suspicion of urethral stricture. The radiation dose of this examination is 5-9 mSV. Sono-urethrography was introduced in 1988 (McAninch et al. , J Urol 1988); the diagnostic accuracy of sono-urethrography is equal compared to conventional urethrography, with even a better measurement of stricture length and degree of spongiofibrosis with sono-urethrography. However, sono-urethrography remained underused among urologists and radiologists.

Patients will be randomly assigned into two groups:

Group A: conventional urethrography Group B: sono-urethrography In case sono-urethrography is inconclusive or of poor quality, a conventional urethrography will be performed.

The radiation dose in the two groups will be measured. The stricture length and location will be recorded and compared with the perioperative findings in order to evaluate the diagnostic accuracy. The complications of the procedure(s) will be recorded with a questionnaire directly after and two weeks after the conventional or sono-urethrography.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a suspicion of urethral stricture disease for which an indication of imaging of the urethra exists.

Exclusion Criteria:

* Transsexual patients.
* Patients with perineostomy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Radiation dose during diagnostic intervention. | During urethrography.
  The radiation dose will be measured with a dosimeter.

SECONDARY OUTCOMES:
Diagnostic accuracy of sono-urethrography vs conventional urethrography. | Immediately and 2 weeks after urethrography
  The results of sono-urethrography and conventional urethrography will be compared with the intraoperative situation (place stricture, length stricture); contrast allergy and complications are scored with a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas Lumen, M.D., Ph.D., Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

REFERENCES:
- See also: Related Info — http://www.uzgent.be